CLINICAL TRIAL: NCT05529394
Title: Effect of Storage Condition on CD47 Expression Level in Platelet Concentrate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abeer Abdallah Ali, Resident doctor, Assiut University
Other Study IDs: Abeer Abdallah Ali
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Platelet Storage Pool Deficiency
MeSH Terms: conditions — Platelet Storage Pool Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Effect of storage condition on CD47 expression level in platelet concentrate

DETAILED DESCRIPTION:
CD47 is a cell surface glycoprotein expressed on all cell types .It is an attractive target for therapy because it is involved in regulation of cell survival and cell death by acting as a ligand for signal-regulatory protein alpha expressed on macrophages

ELIGIBILITY:
Inclusion Criteria:

* donors met AABB criteria

Exclusion Criteria:

* donors not met AABB criteria

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: Effect of storage condition on CD47 expression level in platelet concentrate
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of CD47 expression level on platelets by exposure to different storage temperatures | 3 years
  To increase survival time of platelets